CLINICAL TRIAL: NCT01369589
Title: An Evaluation of the Impact of a Single Dose of P-552 on Oral Mucosal Wetness in Subjects With Xerostomia Related to Sjogren's Syndrome
Brief Title: An Evaluation of the Impact of a Single Dose of P-552 on Oral Mucosal Wetness
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Parion Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 552-209S
Record Dates: First submitted 2011-06-06; First posted 2011-06-09 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-03

CONDITIONS: Xerostomia; Sjogren's Syndrome
Keywords: Xerostomia; dry mouth; Sjogren's Syndrome
MeSH Terms: conditions — Xerostomia; Sjogren's Syndrome | interventions — Water; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- P-552 on Day 1 and Placebo on Day 2 (Experimental): Randomly assigned subjects will receive a single dose of P-552 on Day 1 followed by a single dose of Placebo on Day 2
  Interventions: Drug: P-552; Drug: Placebo
- Placebo on Day 1 and P-552 on Day 2 (Experimental): Randomly assigned subjects will receive a single dose of Placebo on Day 1 followed by a single dose of P-52 on Day 2
  Interventions: Drug: P-552; Drug: Placebo

INTERVENTIONS:
Drug: P-552 — P-552 will be administered as 10 mL mouth rinse to be swished in the mouth fro 30 seconds and then completely expectorated.
  Other Names: P-552 Oral Rinse
Drug: Placebo — Placebo will be administered as 10 mL mouth rinse to be swished in the mouth for 30 seconds and then completely expectorated.
  Other Names: Vehicle Oral Rinse; Water for Injection

SUMMARY:
The primary objective of this clinical study is to determine the impact of P-552 oral rinse on salivary volume after administration of a single dose of P-552and versus vehicle rinse. Changes in oral mucosal wetness will be assessed via collection of salivary output and via measurement of oral wetness using the Periotron 8000 instrument.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged 18 years or older, and who are capable of providing their written informed consent to participate in the study.
2. Male subjects must be either not sexually active, surgically sterilized, or agree to use an appropriate "double-barrier" method (such as a diaphragm and condom) during study participation and for at least 30 days after the completion of dosing.
3. Non-pregnant female subjects must be either not sexually active, postmenopausal, or surgically sterilized; or agree to use an appropriate "double-barrier" method (such as a diaphragm and condom); or are currently using a prescribed transdermal, injection, implant, or oral contraceptive for at least 30 days before receiving the first dose of study drug during study participation and at least 30 days after the completion of dosing.
4. Are in good health, as determined by a medical history, a physical examination, a detailed oral examination, and results of clinical chemistry, hematology and urinalysis.
5. Has minimal level of unstimulated whole mouth salivary flow (greater than or equal to 0.05 milliliters [i.e., 0.05 grams] per 5 minutes) at the screening visit.
6. Have a diagnosis of primary Sjogren's syndrome consistent with the revised version of the European criteria proposed by the American-European Consensus Group European Cooperative Community Classification Criteria for Sjogren's Syndrome.

Exclusion Criteria:

1. Regularly uses antihistamines that have been started or the dose adjusted within the last 30 days.
2. Has started using systemic cholinergic secretagogues or tricyclic antidepressant drugs within 12 weeks before Screening, is not on a stable dosing regimen for at least 14 days prior to the Screening visit, or is unable to maintain stable dosing throughout the study.
3. Is unable to withhold the use of systemic cholinergic secretagogues and oral comfort agents (e.g., OraMoist, MouthKote, Biotene products, etc.) on the morning of each study visit and until 2 hours after dosing at study visits; and is unable to take the last nighttime dose at a standard time throughout the study.
4. Is unable to maintain a stable dosage regimen of any concomitant medication throughout the duration of the trial.
5. Shows evidence of a significant active or ongoing oral infection or other oral conditions (e.g., lichen planus) that, in the opinion of the investigator, might affect the safety of the subject or might exacerbate during study participation.
6. Has acutely infected salivary glands (with or without pain) or suspected closure of the salivary glands.
7. Has received an investigational drug within the past 30 days.
8. Has a history of allergy to any medicine chemically related to the study drug (e.g., amiloride, Moduretic, Midamor, triamterene).
9. Has a present history of any clinically significant and uncontrolled neurologic, gastrointestinal, renal, hepatic, cardiovascular (including hyper/hypotension and tachy/bradycardia), psychological, pulmonary, metabolic, endocrine, or hematological disorder or disease, or any other major disorder or disease, in the opinion of the investigator.
10. Has viral hepatitis or tested positively for the hepatitis B surface antigen or hepatitis C (nonA, non-B) antibody, or a positive result for human immunodeficiency virus antibodies.
11. Has a positive serum pregnancy test or is nursing (female subjects only).
12. Should not participate in the study, in the opinion of the Principal or Clinical investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Salivary volume | 60 minutes
Salivary Volume | 120 minutes

SECONDARY OUTCOMES:
Periotron measurement | 15, 30 and 90 minutes
  measurement of mucosal wetness

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States